CLINICAL TRIAL: NCT00575523
Title: Atropine for Prevention of Dysrhythmias Caused by Percutaneous Ethanol Instillation for Hepatoma Therapy
Acronym: atropinePEI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnulf Ferlitsch, MD, Gastroenterology and Hepatology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: atropinePEI
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Arrhythmia; Respiratory Arrest
Keywords: atropine; percutaneous ethanol instillation; hepatoma; bradycardia; arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac; Apnea; Carcinoma, Hepatocellular; Bradycardia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Atropine (Active Comparator): Atropine 0,5mg is administered intravenously immediately before starting percutaneous ethanol instillation.
  Interventions: Drug: Atropine
- 2: Placebo (Placebo Comparator): 1ml 0,9% Saline solution is administered intravenously immediately before starting percutaneous ethanol instillation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine — Atropine 0,5mg is administered once intravenously immediately before starting percutaneous ethanol instillation.
  Arms: 1: Atropine
Drug: Placebo — 1ml 0,9% Saline solution is administered intravenously immediately before starting percutaneous ethanol instillation.
  Arms: 2: Placebo

SUMMARY:
Ultrasound guided percutaneous ethanol injection (PEI) is an established method in the treatment of hepatocellular carcinoma (HCC) and considered a safe procedure with severe complications occurring rarely. Previous studies revealed, that the occurrence of bradycardia and sinuatrial blockage is quite frequent during ethanol instillation sometimes accompanied by clinical complications such as unconsciousness, respiratory arrest or seizure like symptoms. Study purpose is to evaluate whether the use of i.v. Atropine before starting ethanol instillation can prevent dysrhythmias during instillation. Study design: randomized, placebo controlled, double blinded study. Atropine or saline solution will be administered intravenously to 40 patients immediately before starting percutaneous ethanol instillation. A 6 line ECG with limb leads will be recorded at rest and during ethanol instillation to reveal possibly occurring dysrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatoma scheduled for treatment with percutaneous ethanol instillation

Exclusion Criteria:

* contraindication for the administration of atropine like
* narrow angle glaucoma
* mechanic stenoses of the GI-tract
* clinically relevant prostatic hypertrophy
* paralytic ileus
* myasthenia gravis
* severe cerebral sclerosis
* acute lung edema
* acute myocardial infarction
* cardiac insufficiency
* hyperthyroidism
* patients with contraindication to undergo percutaneous ethanol instillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-10; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of dysrhythmias | during percutaneous ethanol instillation

SECONDARY OUTCOMES:
Clinical complications | during percutaneous ethanol instillation and consecutive 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Div. of Gastroenterology and Hepatology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ferlitsch A, Kreil A, Bauer E, Schmidinger H, Schillinger M, Gangl A, Peck-Radosavljevic M. Bradycardia and sinus arrest during percutaneous ethanol injection therapy for hepatocellular carcinoma. Eur J Clin Invest. 2004 Mar;34(3):218-23. doi: 10.1111/j.1365-2362.2004.01321.x. PMID 15025681
- [Derived] Arnulf F, Monika S, Herwig S, Monika H, Johannes PD, Gregor U, Alfred G, Markus PR. Atropine for prevention of cardiac dysrhythmias in patients with hepatocellular carcinoma undergoing percutaneous ethanol instillation: a randomized, placebo-controlled, double-blind trial. Liver Int. 2009 May;29(5):715-20. doi: 10.1111/j.1478-3231.2008.01905.x. Epub 2008 Oct 27. PMID 19018977